CLINICAL TRIAL: NCT06953700
Title: Effects of Asymmetries on Binaural-Hearing Abilities Across the Lifespan
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1959852; 1R21DC021825 (NIH)
Record Dates: First submitted 2025-04-15; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Aging; Hearing Loss; Hearing Asymmetry
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test of Hearing Function in Acoustic Hearing Listeners (Experimental)
  Interventions: Diagnostic Test: Test of hearing function

INTERVENTIONS:
Diagnostic Test: Test of hearing function — These are measurements of hearing acuity and spatial hearing.

SUMMARY:
Binaural hearing involves combining auditory information across the ears. With binaural hearing, listeners benefit from perceiving sounds from different spatial locations. This is critical in solving the "cocktail party problem" (i.e., understanding speech in the presence of competing background sounds and noise). As humans get older, hearing loss increases, binaural abilities decrease, and the cocktail party problem becomes increasingly difficult. This research studies the mechanisms underlying the impact of age and hearing loss on speech-perception in noise and cocktail-party listening situations. More specifically, the role of hearing asymmetries between the ears is investigated. The specific aims are to generate an audiological and binaural-hearing-focused dataset for a large cohort of participants that vary in hearing asymmetry, age, and hearing loss and to use machine learning to uncover complex associations and generate novel hypotheses relating audiometric variables and basic binaural-hearing abilities to the cocktail-party problem. Participants in this research will complete perceptual measures of hearing acuity and spatial hearing. Participants will also report on speech understanding under noisy and challenging listening conditions. This research may lead to improvements in audiological care and hearing interventions.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-80 years)
* No hearing asymmetry between ears (≤10 dB at any frequency) or, hearing asymmetry between ears >10 dB
* Native English speakers
* Primarily use oral language
* Sufficient corrected or uncorrected visual acuity (20/50 or better) to read large-font text

Exclusion Criteria:

* Acoustic tone-detection threshold >50 dB HL at any octave frequency (250-4000 Hz) in either ear (i.e., more than a moderate hearing loss)
* History of neurological disorders (e.g., stroke, Parkinson's disease) determined by self-report
* History of post-traumatic stress disorder or traumatic brain injury determined by self-report
* Possibility of acoustic neuroma, hearing asymmetry (>10 dB at three consecutive audiometric threshold frequencies)
* Montreal Cognitive Assessment (MoCA) score <22/30
* No oral language use
* Cochlear implant user
* Conductive hearing loss

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Sound localization | After enrollment, in one visit lasting 1-2 hours
  A measure of sound localization ability (summarizing the ability using broadband and narrowband noise stimuli). Localization is the ability to accurately report the location from which a sound source originated. The difference between actual and reported locations is used for the measure. (Units, angle measure in degrees)
Spatial release from masking | After enrollment, in one visit lasting 1-2 hours
  A measure of speech understanding. Spatial release from masking is calculated by finding the difference in thresholds between listening with co-located vs. separated masking signals. (Units, dB)

SECONDARY OUTCOMES:
Basic binaural sensitivity | After enrollment, in one visit lasting 1-2 hours
  A summary measure of basic binaural sensitivity (discrimination thresholds) that uses both frequency-specific and more broadband stimuli that differ in interaural time and level cues. (Units dB)
Cognitive assessment | After enrollment, in one visit lasting 1-2 hours
  A control measurement for factors that may contribute to hearing deficit. The standardized Montreal Cognitive Assessment cognitive screener and NIH Toolbox subscores for Working Memory, Processing Speed, and Attention will be combined to summarize a potential cognitive contribution to hearing deficits. (Units, points.)
Audiological assessment of hearing thresholds | After enrollment, in one visit lasting ~1 hour
  Measurement of hearing thresholds by presenting sounds of specific frequencies via audiometer and recording the lowest level that can be detected for each frequency. These thresholds are then averaged. (Units, dB)
Auditory Brainstem Response | After enrollment, in one visit lasting ~1 hour
  A non-invasive measure of auditory processing integrity past the point of the cochlea. Earphones are used to present brief acoustic click stimuli and waveform recordings of neural activity at the level of the brainstem are collected via surface sensors on the listener's head. (Unit, latency in milliseconds)
Distortion-Product Otoacoustic Emissions | After enrollment, in one visit lasting ~1 hour
  A measurement of the inner ear's acoustic response to a brief stimulus played in the ear canal. This can provide information about the integrity of the cochlea's outer hair cells. (Units, dB SNR (signal to noise ratio))

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Goupell, PhD, Principal Investigator — University of Maryland, College Park; Michael P. Cummings, PhD, Study Director — University of Maryland, College Park
Locations (1):
- University of Maryland, College Park, College Park, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data that document, support, and validate research findings will be made available when the main findings have been accepted for publication. De-identified data relevant to the project will be disseminated to researchers on and off-campus by request and review of the PI.
  After publication, research products from this project will be archived at the Digital Repository at the University of Maryland (DRUM) (unless a more appropriate facility can be identified). DRUM is a long-term, open access repository managed and maintained by the University of Maryland Libraries. Researchers and the general public can download data and code files, associated metadata and documentation, and any guidelines for reuse.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following publication, available for at least seven years.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee.